CLINICAL TRIAL: NCT01761279
Title: A Prospective Single-blind Observational Cohort Study of High Definition White Light Endoscopy and i-Scan Image Enhancement for the Characterisation of Small Colonic Polyps
Brief Title: High Definition Endoscopy With i-Scan for Small Colonic Polyp Evaluation: The HiScope Study
Acronym: HiSCOPE
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Pradeep Bhandari, Professor of Gastroenterology, Portsmouth Hospitals NHS Trust
Other Study IDs: PHT/2009/046
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Colonic Polyps
Keywords: Colonic polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: High definition white light endoscopy

SUMMARY:
Current standard practice is to remove all colonic polyps found during colonoscopy as it has not been possible to distinguish between polyps with some malignant potential (adenomatous) and those with negligable malignant potential (non-adenomatous).

Recent advances in endoscope imaging and technology have allowed endoscopists to distinguish between these two types of polyps by examining minute surface details.

i-Scan is a new digital enhancement method that aims to enhance surface details and may enable similar accurate distinction between adenomatous and non-adenomatous polyps.

Hypothesis:

High definition white light endoscopy plus i-Scan improves diagnostic accuracy of in-vivo assessment of colonic polyps <10mm in size over high definition white light endoscopy alone.

DETAILED DESCRIPTION:
Traditionally all polyps detected at colonoscopy, except obvious cancers, have been removed. It is felt that small (<10mm diameter) hyperplastic polyps cannot be reliably distinguished from adenomatous polyps by endoscopists [1]. Therefore a large number of hyperplastic polyps are removed unnecessarily. This results in increased risk to patients through exposing them to unnecessary polypectomy, and increased cost to the health service through the cost of processing greater numbers of histopathology specimens. The cost per specimen is around £58.

This challenge of distinguishing small hyperplastic polyps from small adenomatous polyps has been met over the past decade through the use of novel chromoendoscopy and computed 'virtual chromoendoscopy' techniques.

Chromoendoscopy involves using staining or contrast dyes to highlight the minute surface patterns in the mucosa of the gastrointestinal tract. The dyes are applied to the colonic mucosa via the working channels of the endoscope. Vital stains such as cresyl violet and methylene blue, which are taken up into epithelial cells, have been used by Japanese endoscopists for many years. Work by Kudo et al showed that by using these stains in combination with magnification endoscopy the minute 'pit patterns' of colonic mucosal lesions could be precisely examined and classified. The pits described are the surface opening of the mucosal crypts. Kudo showed that the surface pit pattern could predict the histology of a lesion with high accuracy [2-4], enabling distinction between adenomatous and hyperplastic polyps. Concerns regarding potential harmful effects of vital stains increased the popularity of an alternative chromoendoscopy dye, indigocarmine [5]. Indigocarmine is not taken up by cells but lies on the colonic wall. Studies from East Asia, the USA and Europe published in the early part of the last decade showed that by combining indigocarmine and magnification endoscopy, neoplastic colonic polyps (adenomas) could be distinguished from non-neoplastic hyperplastic polyps with accuracy rates of 68-96% [6-10]. By the same method, surface patterns could also identify small early colorectal cancers[11] . Subsequent studies demonstrated that indigocarmine could adequately distinguish between adenomatous and hyperplastic polyps without the need for optical magnification [12-15].

During the past few years new methods of closely examining lesions within the colon have been developed. Digital imaging techniques or 'virtual chromoendoscopy' systems have been developed by endoscope manufacturers as a 'push-button' alternative to chromoendoscopy dyes, being potentially simpler and quicker to use. The first of these novel technologies available was the narrow band imaging (NBI) system produced by Olympus. A filter within the endoscope selects out narrow bandwidths of blue and green light, and thus reduces red light. These wavelengths penetrate only the superficial layers of the mucosa, highlighting surface patterns and microvasculature. Adenomatous polyps have more numerous and prominent microvessels in comparison to hyperplastic poylps. This system has been shown to be effective in differentiating small hyperplastic and adenomatous polyps with accuracies of 91 - 94% [16-23].

The Fujinon Intelligent Colour Enhancement (FICE) system developed by Fujinon uses post-processor electronic colour filter technology to allow a range of filter images with different wavelengths of light to be viewed. Similar results to NBI have been achieved in the characterisation of small polyps [13, 24, 25].

More recently a further virtual chromoendoscopy system, i-Scan has been developed by Pentax. i-Scan identifies areas of contrast between adjacent pixels (ie light bordering dark) and enhances this contrast. Additionally in a similar method to FICE, post-processor manipulation of the red, green and blue components of the spectrum is used to enhance vessels and surface structures.

A single study from Germany has suggested that i-Scan improves the detection of lesions during flexible sigmoidoscopy and can accurately predict histology. There is a need for further data on the clinical efficacy of i-Scan in the assessment of colonic polyps, particularly in a UK population and in a bowel cancer screening population, neither of which have been studied to date.

Through the use of these new technologies it may be possible to accurately predict the histology of small polyps in real time. Once an in-vivo diagnosis has been made with high confidence it may be possible for small hyperplastic polyps to be discarded, rather than sent for histological analysis, or to be left in situ [22]. This has potential benefits in reducing the frequency and consequent risk of polypectomy for patients and could also reduce pathology costs. UK and US guidelines for repeat surveillance colonoscopy after adenomas are detected at baseline examination are based on the number and size and histology of adenomas [26, 27]. At present these 'rescope intervals' are determined once the histology report of any resected polyps is received. With accurate in-vivo diagnosis these intervals may be set immediately after the baseline colonoscopy has been completed.

Whilst the development of these endoscopic advanced imaging technologies is to be welcomed, it is important for studies to determine what can be achieved through their use, over and above standard white-light colonoscopy. The American Society for Gastrointestinal Endoscopy has identified the utility of technologies used in the real-time assessment of diminutive (<5mm) colonic polyps as a key area for study, and has published guidelines on the minimum standards which new endoscopic technologies should meet before their use becomes widely adopted [28].

We aim to evaluate HDWL and HDWL + i-Scan for the real time assessment and prediction of histology of small colonic polyps in a BCSP population.

ELIGIBILITY:
Inclusion Criteria:

* Patients found to have colonic polyps up to 10mm in size

Exclusion Criteria:

* Poor bowel preparation
* Inflammatory bowel disease
* Polyposis syndrome

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK Bowel Cancer Screening patients attending for colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MBBS, Principal Investigator — Portsmouth Hospitals NHS Trust

REFERENCES:
- [Background] Norfleet RG, Ryan ME, Wyman JB. Adenomatous and hyperplastic polyps cannot be reliably distinguished by their appearance through the fiberoptic sigmoidoscope. Dig Dis Sci. 1988 Sep;33(9):1175-7. doi: 10.1007/BF01535796. PMID 3044716
- [Background] Kudo S, Hirota S, Nakajima T, Hosobe S, Kusaka H, Kobayashi T, Himori M, Yagyuu A. Colorectal tumours and pit pattern. J Clin Pathol. 1994 Oct;47(10):880-5. doi: 10.1136/jcp.47.10.880. PMID 7962600
- [Background] Kudo S, Rubio CA, Teixeira CR, Kashida H, Kogure E. Pit pattern in colorectal neoplasia: endoscopic magnifying view. Endoscopy. 2001 Apr;33(4):367-73. doi: 10.1055/s-2004-826104. No abstract available. PMID 11315901
- [Background] Kudo S, Tamura S, Nakajima T, Yamano H, Kusaka H, Watanabe H. Diagnosis of colorectal tumorous lesions by magnifying endoscopy. Gastrointest Endosc. 1996 Jul;44(1):8-14. doi: 10.1016/s0016-5107(96)70222-5. PMID 8836710
- [Background] Davies J, Burke D, Olliver JR, Hardie LJ, Wild CP, Routledge MN. Methylene blue but not indigo carmine causes DNA damage to colonocytes in vitro and in vivo at concentrations used in clinical chromoendoscopy. Gut. 2007 Jan;56(1):155-6. doi: 10.1136/gut.2006.107300. No abstract available. PMID 17172595
- [Background] De Palma GD, Rega M, Masone S, Persico M, Siciliano S, Addeo P, Persico G. Conventional colonoscopy and magnified chromoendoscopy for the endoscopic histological prediction of diminutive colorectal polyps: a single operator study. World J Gastroenterol. 2006 Apr 21;12(15):2402-5. doi: 10.3748/wjg.v12.i15.2402. PMID 16688833
- [Background] Eisen GM, Kim CY, Fleischer DE, Kozarek RA, Carr-Locke DL, Li TC, Gostout CJ, Heller SJ, Montgomery EA, Al-Kawas FH, Lewis JH, Benjamin SB. High-resolution chromoendoscopy for classifying colonic polyps: a multicenter study. Gastrointest Endosc. 2002 May;55(6):687-94. doi: 10.1067/mge.2002.123619. PMID 11979251
- [Background] Fu KI, Sano Y, Kato S, Fujii T, Nagashima F, Yoshino T, Okuno T, Yoshida S, Fujimori T. Chromoendoscopy using indigo carmine dye spraying with magnifying observation is the most reliable method for differential diagnosis between non-neoplastic and neoplastic colorectal lesions: a prospective study. Endoscopy. 2004 Dec;36(12):1089-93. doi: 10.1055/s-2004-826039. PMID 15578300
- [Background] Konishi K, Kaneko K, Kurahashi T, Yamamoto T, Kushima M, Kanda A, Tajiri H, Mitamura K. A comparison of magnifying and nonmagnifying colonoscopy for diagnosis of colorectal polyps: A prospective study. Gastrointest Endosc. 2003 Jan;57(1):48-53. doi: 10.1067/mge.2003.31. PMID 12518130
- [Background] Tung SY, Wu CS, Su MY. Magnifying colonoscopy in differentiating neoplastic from nonneoplastic colorectal lesions. Am J Gastroenterol. 2001 Sep;96(9):2628-32. doi: 10.1111/j.1572-0241.2001.04120.x. PMID 11569686
- [Background] Kato S, Fujii T, Koba I, Sano Y, Fu KI, Parra-Blanco A, Tajiri H, Yoshida S, Rembacken B. Assessment of colorectal lesions using magnifying colonoscopy and mucosal dye spraying: can significant lesions be distinguished? Endoscopy. 2001 Apr;33(4):306-10. doi: 10.1055/s-2001-13700. PMID 11315890
- [Background] Sonwalkar S, Rotimi O, Rembacken BJ. Characterization of colonic polyps at conventional (nonmagnifying) colonoscopy after spraying with 0.2 % indigo carmine dye. Endoscopy. 2006 Dec;38(12):1218-23. doi: 10.1055/s-2006-944787. PMID 17163322
- [Background] Pohl J, Lotterer E, Balzer C, Sackmann M, Schmidt KD, Gossner L, Schaab C, Frieling T, Medve M, Mayer G, Nguyen-Tat M, Ell C. Computed virtual chromoendoscopy versus standard colonoscopy with targeted indigocarmine chromoscopy: a randomised multicentre trial. Gut. 2009 Jan;58(1):73-8. doi: 10.1136/gut.2008.153601. Epub 2008 Oct 6. PMID 18838485
- [Background] Su MY, Hsu CM, Ho YP, Chen PC, Lin CJ, Chiu CT. Comparative study of conventional colonoscopy, chromoendoscopy, and narrow-band imaging systems in differential diagnosis of neoplastic and nonneoplastic colonic polyps. Am J Gastroenterol. 2006 Dec;101(12):2711-6. doi: 10.1111/j.1572-0241.2006.00932.x. PMID 17227517
- [Background] Apel D, Jakobs R, Schilling D, Weickert U, Teichmann J, Bohrer MH, Riemann JF. Accuracy of high-resolution chromoendoscopy in prediction of histologic findings in diminutive lesions of the rectosigmoid. Gastrointest Endosc. 2006 May;63(6):824-8. doi: 10.1016/j.gie.2005.09.013. PMID 16650546
- [Background] East JE, Suzuki N, Bassett P, Stavrinidis M, Thomas HJ, Guenther T, Tekkis PP, Saunders BP. Narrow band imaging with magnification for the characterization of small and diminutive colonic polyps: pit pattern and vascular pattern intensity. Endoscopy. 2008 Oct;40(10):811-7. doi: 10.1055/s-2008-1077586. Epub 2008 Sep 30. PMID 18828077
- [Background] Henry ZH, Yeaton P, Shami VM, Kahaleh M, Patrie JT, Cox DG, Peura DA, Emura F, Wang AY. Meshed capillary vessels found on narrow-band imaging without optical magnification effectively identifies colorectal neoplasia: a North American validation of the Japanese experience. Gastrointest Endosc. 2010 Jul;72(1):118-26. doi: 10.1016/j.gie.2010.01.048. Epub 2010 Apr 9. PMID 20381799
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Background] Rastogi A, Keighley J, Singh V, Callahan P, Bansal A, Wani S, Sharma P. High accuracy of narrow band imaging without magnification for the real-time characterization of polyp histology and its comparison with high-definition white light colonoscopy: a prospective study. Am J Gastroenterol. 2009 Oct;104(10):2422-30. doi: 10.1038/ajg.2009.403. Epub 2009 Jul 7. PMID 19584829
- [Background] Rastogi A, Bansal A, Wani S, Callahan P, McGregor DH, Cherian R, Sharma P. Narrow-band imaging colonoscopy--a pilot feasibility study for the detection of polyps and correlation of surface patterns with polyp histologic diagnosis. Gastrointest Endosc. 2008 Feb;67(2):280-6. doi: 10.1016/j.gie.2007.07.036. Epub 2007 Dec 26. PMID 18155210
- [Background] Rogart JN, Jain D, Siddiqui UD, Oren T, Lim J, Jamidar P, Aslanian H. Narrow-band imaging without high magnification to differentiate polyps during real-time colonoscopy: improvement with experience. Gastrointest Endosc. 2008 Dec;68(6):1136-45. doi: 10.1016/j.gie.2008.04.035. Epub 2008 Aug 8. PMID 18691708
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] Hoffman A, Kagel C, Goetz M, Tresch A, Mudter J, Biesterfeld S, Galle PR, Neurath MF, Kiesslich R. Recognition and characterization of small colonic neoplasia with high-definition colonoscopy using i-Scan is as precise as chromoendoscopy. Dig Liver Dis. 2010 Jan;42(1):45-50. doi: 10.1016/j.dld.2009.04.005. Epub 2009 May 26. PMID 19473893
- [Background] Teixeira CR, Torresini RS, Canali C, Figueiredo LF, Mucenic M, Pereira Lima JC, Carballo MT, Saul C, Toneloto EB. Endoscopic classification of the capillary-vessel pattern of colorectal lesions by spectral estimation technology and magnifying zoom imaging. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):750-6. doi: 10.1016/j.gie.2008.09.062. PMID 19251021
- [Background] Togashi K, Osawa H, Koinuma K, Hayashi Y, Miyata T, Sunada K, Nokubi M, Horie H, Yamamoto H. A comparison of conventional endoscopy, chromoendoscopy, and the optimal-band imaging system for the differentiation of neoplastic and non-neoplastic colonic polyps. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):734-41. doi: 10.1016/j.gie.2008.10.063. PMID 19251019
- [Background] Cairns S, Scholefield JH. Guidelines for colorectal cancer screening in high risk groups. Gut. 2002 Oct;51 Suppl 5(Suppl 5):V1-2. doi: 10.1136/gut.51.suppl_5.v1. PMID 12221029
- [Background] Levin B, Lieberman DA, McFarland B, Smith RA, Brooks D, Andrews KS, Dash C, Giardiello FM, Glick S, Levin TR, Pickhardt P, Rex DK, Thorson A, Winawer SJ; American Cancer Society Colorectal Cancer Advisory Group; US Multi-Society Task Force; American College of Radiology Colon Cancer Committee. Screening and surveillance for the early detection of colorectal cancer and adenomatous polyps, 2008: a joint guideline from the American Cancer Society, the US Multi-Society Task Force on Colorectal Cancer, and the American College of Radiology. CA Cancer J Clin. 2008 May-Jun;58(3):130-60. doi: 10.3322/CA.2007.0018. Epub 2008 Mar 5. PMID 18322143
- [Background] Rex DK, Kahi C, O'Brien M, Levin TR, Pohl H, Rastogi A, Burgart L, Imperiale T, Ladabaum U, Cohen J, Lieberman DA. The American Society for Gastrointestinal Endoscopy PIVI (Preservation and Incorporation of Valuable Endoscopic Innovations) on real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2011 Mar;73(3):419-22. doi: 10.1016/j.gie.2011.01.023. PMID 21353837
- [Derived] Basford PJ, Longcroft-Wheaton G, Higgins B, Bhandari P. High-definition endoscopy with i-Scan for evaluation of small colon polyps: the HiSCOPE study. Gastrointest Endosc. 2014 Jan;79(1):111-8. doi: 10.1016/j.gie.2013.06.013. Epub 2013 Jul 17. PMID 23871094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients attending for colonoscopy at Portsmouth Hospitals NHS Trust throught the Bowel Cancer Screening programme were recruited from May 2010-May 2011.
Pre-assignment Details: Cohort study - single cohort. Patients found to have inflammatory bowel disease or a polyposis syndrome were excluded
Groups:
- HDWL and i-Scan Assessment: High Definition White Light Endoscopy.
Period: Overall Study
Arm/Group | HDWL and i-Scan Assessment
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HDWL + I-Scan: High Definition White Light Endoscopy and i-Scan assessment performed of all polyps
Arm/Group | HDWL + I-Scan
Number analyzed (Participants) | 84
Age Continuous [Mean (Full Range); unit: Years] | 67.6 [60 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of In-vivo Polyp Assessment
Description: Diagnostic accuracy of in-vivo assessment of colonic polyps <10mm in size using high definition white light endoscopy and high definition white light endoscopy plus i-Scan image enhancement. Accuracy compared to the gold standard of histopathology. Accuracy - number of polyps with histology correctly predicted by in-vivo method/total number of polyps assessed (Expressed as a percentage)
Time Frame: Once histopathology results are known, approximately 2 weeks after in-vivo assessment
Population: There were 84 patients included in the study. 209 polyps <10mm included in the study.
Measure: Number (95% Confidence Interval); unit: % diagnostic accuracy
Units Other Than Participants: Polyps <10mm in size
Groups:
- HDWL: High Definition White Light Endoscopy
- i-Scan: High definition white light endoscopy with i-Scan image enhancement
Arm/Group | HDWL | i-Scan
Number analyzed (Participants) | 84 | 84
Number analyzed (Polyps <10mm in size) | 209 | 209
% diagnostic accuracy | 93.3 [88.5 to 96.3] | 94.7 [90.3 to 97.2]

2. Secondary Outcome: Sensitivity for Adenomatous Histology of Colonic Polyps <10mm in Size
Description: Sensitivity for adenomatous histology of in-vivo assessment of colonic polyps <10mm in size using high definition white light endoscopy and high definition white light endoscopy plus i-Scan image enhancement. Sensitivity compared to the gold standard of histopathology. Senstivity for adenomatous histology = number of correctly identified adenomas (true positives)/total number of adenomas (true positives + false negatives)
Time Frame: Once histopathology results are known, approximately 2 weeks after in-vivo assessment
Population: 134 is the number of adenomatous polyps included in the study.
Measure: Number (95% Confidence Interval); unit: Percentage sensitivity
Units Other Than Participants: Adenomatous polyps <10mm in size
Arm/Group | HDWL | i-Scan
Number analyzed (Participants) | 84 | 84
Number analyzed (Adenomatous polyps <10mm in size) | 134 | 134
Percentage sensitivity | 95.5 [91.8 to 97.8] | 97.0 [93.6 to 98.9]

3. Secondary Outcome: Specificity for Adenomatous Histology of Colonic Polyps <10mm in Size
Description: Specificity for adenomatous histology of in-vivo assessment of colonic polyps <10mm in size using high definition white light endoscopy and high definition white light endoscopy plus i-Scan image enhancement. Specificity compared to the gold standard of histopathology. Specificity for adenomatous histology = number of correctly identified non-neoplastic polyps (true negatives)/total number of non-neoplastic polyps (true negatives + false positives)
Time Frame: Once histopathology results are known, approximately 2 weeks after in-vivo assessment
Population: 75 is the number of non-neoplastic polyps included in the study.
Measure: Number (95% Confidence Interval); unit: Percentage specificity
Units Other Than Participants: Non-neoplastic polyps <10mm in size
Arm/Group | HDWL | i-Scan
Number analyzed (Participants) | 84 | 84
Number analyzed (Non-neoplastic polyps <10mm in size) | 75 | 75
Percentage specificity | 89.3 [82.7 to 93.5] | 90.7 [84.5 to 94.0]

4. Secondary Outcome: Negative Predictive Value for Adenomatous Histology of Rectosigmoid Polyps ≤5mm in Size
Description: Negative predictive value for adenomatous histology of rectosigmoid polyps ≤5mm in size using high definition white light endoscopy and high definition white light endoscopy plus i-Scan image enhancement. NPV compared to the gold standard of histopathology. Negative predictive value = number of true negatives/(number of true negatives + number of false negatives)
Time Frame: Once histopathology results are known, approximately 2 weeks after in-vivo assessment
Population: Numbers indicate the number of rectosigmoid polyps <5mm in size assessed as being non-neoplastic
Measure: Number (95% Confidence Interval); unit: Percentage Negative Predictive Value
Units Other Than Participants: Rectosigmoid Polyps <5mm
Arm/Group | HDWL | i-Scan
Number analyzed (Participants) | 84 | 84
Number analyzed (Rectosigmoid Polyps <5mm) | 46 | 48
Percentage Negative Predictive Value | 100 [92.8 to 100] | 100 [93.4 to 100]

5. Other Pre Specified Outcome: Accuracy of Prediction of Polyp Surveillence Intervals
Description: Accuracy of prediction of post-polypectomy surveillence colonoscopy intervasl based on national guidelines. Intervals based on in-vivo assessment of all polyps ≤5mm in size combined with histopathology of polyps >5mm in size will be compared to intervals determined by histopathology of all polyps
Time Frame: Once histopathology results are known, approximately 2 weeks after in-vivo assessment
Population: 84 study participants in total. One patient excluded from this analysis as a single polyp was not retrieved for histological analysis.
Measure: Number; unit: Percentage correct surveillence interval
Arm/Group | HDWL | i-Scan
Number analyzed (Participants) | 83 | 83
Percentage correct surveillence interval | 95.3 | 97.2

ADVERSE EVENTS:
Arm/Group | HDWL + I-Scan
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 0/84

LIMITATIONS AND CAVEATS:
Single centre study. Single endoscopist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes